CLINICAL TRIAL: NCT04375033
Title: CSP #2014 - Comparative Effectiveness of Two Formulations of Buprenorphine for Treating Opioid Use Disorder in Veterans (VA-BRAVE)
Brief Title: A Study Comparing Oral Buprenorphine and Injectable Buprenorphine for the Treatment of Opioid Use Disorder
Acronym: VA-BRAVE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014
Record Dates: First submitted 2020-04-03; First posted 2020-05-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
Keywords: Buprenorphine; Veterans; Clinical Trial; Opioid Abstinence; Retention in Care; Pharmacotherapy
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naloxone

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 and assigned to receive at each 28-day research visit either: 1) a 28-day take-home supply of SL buprenorphine, prescribed at the clinically determined dose, or 2) injectable sub-cutaneous buprenorphine administered in the clinic (target dose = 300mg; 100mg dose may be used for those who cannot tolerate 300mg).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sublingual Arm (Experimental): The sublingual buprenorphine contains naloxone in a ratio of 4:1 and will be prescribed. Consistent with the SAMHSA guidelines, before SL-BUP/NLX is prescribed, participants will be evaluated for recent (within 24 hours) drug use and associated symptoms.
  The randomization dose will be determined based on the maintenance dose identified during the induction period, with a target dose of 4-32mg that is standard practice. While the target dose is 4-32mg, occasionally patients may prefer lower doses. SL-BUP/NLX will be prescribed at the randomization visit (28-day supply), then every 4 weeks through week 48.
  Interventions: Drug: Sublingual buprenorphine with naloxone
- Injectable Arm (Experimental): Injectable buprenorphine consists of a depot injectable formulation in polymeric solution and releases buprenorphine over a 28-day (4-week) period by diffusion as the polymer biodegrades. The injection will be administered subcutaneously at each 28-day visit. The target dose is 300mg, there is the option to use 100mg dose. The final study dose of injectable buprenorphine will be given at Week 48.
  Interventions: Drug: Injectable subcutaneous buprenorphine

INTERVENTIONS:
Drug: Sublingual buprenorphine with naloxone — The combination SL-containing buprenorphine contains naloxone in a ratio of 4:1 buprenorphine:naloxone. Participants will be given a 28-prescription at each 28-day visit through Week 48.
  Arms: Sublingual Arm
Drug: Injectable subcutaneous buprenorphine — Injectable buprenorphine consists of a depot injectable formulation in polymeric solution and releases buprenorphine over a 28-day (4-week) period by diffusion as the polymer biodegrades. The injection will be administered subcutaneously at each 28-day visit through Week 48.
  Arms: Injectable Arm

SUMMARY:
VA-BRAVE will determine whether a 28-day long-acting injectable sub-cutaneous formulation of buprenorphine at a target dose of 300mg is superior in retaining Veterans in opioid treatment and in sustaining opioid abstinence compared to the daily sublingual (under the tongue) buprenorphine formulation at a target dose of 4-32 mg (standard of care). This is an open-label, randomized, controlled trial including 952 Veterans with opioid use disorder (OUD) recruited over 7 years and followed actively for 52 weeks. There are a number of secondary objectives that will be studied as well and include: comorbid substance use, both non-fatal and fatal opioid overdose, HIV and Hepatitis B (HBV) and C (HCV) testing results and risk behaviors, incarceration, quality of life, psychiatric symptoms of depression and posttraumatic stress disorder, housing status, dental health and utilization, and cost-effectiveness.

DETAILED DESCRIPTION:
CSP2014 is the first direct long-term comparison of monthly injectable versus daily SL buprenorphine. In addition to its impact on the care of Veterans, the results of VA-BRAVE will provide critical data to guide effective treatment of opioid use disorder throughout the United States.

The CSP2014 study population is Veterans aged 18 years diagnosed with moderate to severe opioid use disorder (OUD) by Diagnostic and Statistical Manual (DSM)-5th edition criteria. Veterans must be entering a new episode of opioid use disorder care prior to study start.

There are two primary outcomes that address key Veterans Health Administration (VHA) clinical issues related to opioid use disorder treatment. The first is retention on protocol-directed medication treatment (sublingual or injectable sub-cutaneous buprenorphine). The second primary outcome is opioid abstinence using the systematic Timeline Followback method of self-report and corresponding urine toxicology screens.

VA-BRAVE includes a 52-week intervention with multiple study visits and up to a 10-year passive follow-up for the duration of the study. Participants are inducted on daily SL buprenorphine using SAMHSA guidelines and dosed upward for a target dose of 4-32 mg for 1 day (should not exceed 45 days). Once target dose reached, participants are randomized 1:1 and assigned to receive at each 28-day research visit either: 1) a 28-day take-home supply of SL buprenorphine, prescribed at the clinically determined dose, or 2) injectable sub-cutaneous buprenorphine administered in the clinic (target dose = 300mg; 100mg dose may be used for those who cannot tolerate 300mg). Participants also receive Medication Management intervention at these visits.

Study visits for all participants occur at Weeks 1, 2, 3 and 4 post-randomization, and biweekly thereafter through Week 52. Self-reported abstinence and urine toxicology screens are obtained at biweekly visits. Following one year of active follow-up, administrative data will be used to follow participants for up to 10 years for early enrollees and up to 7 years for late enrollees. The recruitment expectation is 7 new participants per study year per study site. There will be up to 20 participating VA Medical Center sites.

ELIGIBILITY:
Inclusion Criteria:

* Has used opioids within 30 days prior to consent or within 30 days prior to entry into a supervised setting -- e.g., opioid use within the 30 days prior to recent (<30 days) incarceration, entry into a detoxification facility, or entry into an inpatient hospital setting
* Have started or are in the process of starting on MOUD via clinical induction on SL-BUP/NLX
* Meets DSM-5 criteria for moderate to severe OUD based on the Mini-International Neuropsychiatric Interview
* Referred to/seeking treatment for OUD and willing to accept "partial-agonist-based" therapy

Exclusion Criteria:

* Is a Veteran less than 18 years of age
* For Veterans of childbearing potential (a premenopausal person capable of becoming pregnant), pregnancy, breastfeeding, and/or failure to practice an effective method of birth control
* Failure to reach maintenance dose of 4mg - 32mg SL-BUP/NLX in 45 days or less.
* Taking a form of prescribed maintenance MOUD (e.g., methadone, buprenorphine or XR-NTX) continuously >45 days prior to randomization
* Has a history of significant adverse effects from buprenorphine and/or naloxone
* Has experienced (within the past 2 weeks) recent suicidal or homicidal ideation that requires acute treatment or hospitalization.
* Is unwilling or unable to provide consent
* Meets criteria for current (past month) DSM-5 severe sedative hypnotic use disorder based on the MINI SHUD module
* Anuria and/or dialysis
* Current moderate to severe COVID-19 symptoms with a risk of intubation or critical illness.
* Medical, psychiatric, behavioral, or logistical condition which, in the judgement of the Local Site Investigator (LSI) or Co-Investigator (Co-I), requires a higher level of acute care and/or makes it unlikely the patient can participate in or complete the 52-week active phase of the study.
* Is actively participating in an interventional clinical trial for which a waiver of dual-enrollment with CSP #2014 has not been obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Retention in Treatment Change | Approximately every 4 weeks until the first period of missed prescription medication coverage lasting at least 4 weeks through week 52
  Measured by receipt of prescribed study drug (via prescription or admission) and assessed via local study team records. Retention-in-treatment is a highly sensitive indicator of effective treatment as discontinuation is strongly associated with recurrence of use to opioids and risk for accidental drug poisoning.
Opioid Abstinence | Approximately every 2 weeks through 52 weeks (active phase) and via EMR review for up to 10 years (passive phase)
  Measured by Timeline Followback (self-report measure of substance use) and urine toxicology free of opioids. Both Timeline Followback and urine toxicology must indicate non-use to indicate abstinence.

SECONDARY OUTCOMES:
Accidental Opioid Poisoning (overdose) | Approximately every 2 weeks through 52 weeks (active phase) and via EMR review for up to 10 years (passive phase)
  Self-reported non-fatal accidental opioid poisoning, hospital records, and CDC data on fatal accidental drug poisoning (by state) will be used to indicate fatal and non-fatal accidental opioid poisoning.
Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) seroconversion | Assessed at baseline, week 24, week 52 (active phase) and via EMR review for up to 10 years (passive phase)
  Assessment will indicate positive seroconversion for HIV, HBV, or HCV based on HIV-1 p24 antigen/antibody with reflex HIV RNA viral load, HBV sAB, sAG with reflex HBV viral load if HBV sAG positive only, and HCV AB with reflex HCV viral load. These tests are recommended as standard care for Veterans with OUD.
Healthcare and Service Utilization | Assess from baseline approximately every 4 weeks through 52 weeks (active phase) and via EMR review for up to 10 years (passive phase)
  An indicator of healthcare and service utilization will be obtained using the Service Utilization Review Form (SURF) that assesses utilization of VHA inpatient and outpatient care clinics, SUD clinics, detoxification programs, and pharmacies located within the VHA and local hospitals. Participants' use of other treatments will be documented on the SURF; non-VA health services will also be captured using the SURF.
Other Addictive Substances | Approximately every 2 weeks through 52 weeks (active phase) and via EMR review for up to 10 years (passive phase)
  Measured by Timeline Followback (self-report measure of substance use) and urine toxicology free of other addictive substances. Both Timeline Followback and urine toxicology must indicate non-use to indicate abstinence.
Opioid Craving | Approximately every 4 weeks through 52 weeks (active phase)
  Opioid craving will be measured on a 10-point Likert scale in response to the question "Please indicate how much you are craving opioids right now."
HIV Sexual and Injection Risk Behaviors | Assessed at baseline, weeks 12, 24, 36, and 52
  HIV sexual and injection risk behaviors will be assessed using NIDA's HIV Risk Behavior tool.
Patient Health Questionnaire (PHQ-9) | Assessed at baseline, weeks 12, 24, 36, and 52
  A measure of depressive symptoms (overall) and suicidality (item 9)
PTSD Checklist for DSM-5 | Assessed at baseline, weeks 12, 24, 36, and 52
  A measure of PTSD symptoms
Texas Christian University Criminal Justice Form | Assessed at baseline, weeks 12, 24, 36, and 52
  A measure of incarceration, arrests, criminal activity.
Dental Quality of Life Questionnaire | Assessed at baseline, weeks 24 and 52
  Self-report measure assessing oral/dental health and quality of life, salivary function, access to and use of dental healthcare.

CONTACTS AND LOCATIONS:
Overall Officials: Ismene L. Petrakis, MD, Study Chair — VA Connecticut Healthcare System West Haven Campus, West Haven, CT; Sandra Ann Springer, MD, Study Chair — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (25):
- United States (25):
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - Phoenix VA Health Care System, Phoenix, AZ, Phoenix, Arizona
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - CERC (VISN1, West Haven, CT), West Haven, Connecticut
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Wilmington VA Medical Center, Wilmington, DE, Wilmington, Delaware
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Dayton VA Medical Center, Dayton, OH, Dayton, Ohio
  - Philadelphia MultiService Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont
  - Hampton VA Medical Center, Hampton, VA, Hampton, Virginia
  - Salem VA Medical Center, Salem, VA, Salem, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - Huntington VA Medical Center, Huntington, WV, Huntington, West Virginia
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petrakis I, Springer SA, Davis C, Ralevski E, Gu L, Lew R, Hermos J, Nuite M, Gordon AJ, Kosten TR, Nunes EV, Rosenheck R, Saxon AJ, Swift R, Goldberg A, Ringer R, Ferguson R. Rationale, design and methods of VA-BRAVE: a randomized comparative effectiveness trial of two formulations of buprenorphine for treatment of opioid use disorder in veterans. Addict Sci Clin Pract. 2022 Jan 31;17(1):6. doi: 10.1186/s13722-022-00286-6. PMID 35101115